CLINICAL TRIAL: NCT02755259
Title: Acute Hemodynamic Effect of Acetazolamide in Pulmonary Hypertension
Acronym: AcuteAZA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH-2016-00089
Record Dates: First submitted 2016-03-24; First posted 2016-04-28 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hypertension, Pulmonary
Keywords: Acetazolamide; Hemodynamics
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetazolamide (Experimental): Diamox 500mg i.v. (1x)
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo Saline injection (1x)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: Placebo
  Arms: Placebo

SUMMARY:
To study the acute effect of acetazolamide (AZA) on pulmonary hemodynamics in patients with pulmonary hypertension (PH) undergoing clinically indicated right heart catheterisation (RHC).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) of various etiologies causes dyspnea, impairs exercise performance and is associated with reduced quality of life (QoL) and survival. Treatment options include therapy for any underlying causes, pulmonary vasodilator drugs, oxygen and, in selected cases, pulmonary endarterectomy or lung transplantation. Unfortunately, PH specific drugs are expensive, associated with side effects and even combined pharmacological treatment is often not sufficient to achieve clinical benefits. Therefore, novel therapeutic drugs are needed. The investigators have recently demonstrated that sleep related breathing disorders, which are common in PH patients, can be improved by both nocturnal oxygen therapy and acetazolamide (AZA). AZA is a carbonic anhydrase (CA) inhibitor that acts as a respiratory stimulant thereby improving oxygenation and possibly PH. There are even data suggesting that CA-inhibitors have a direct pulmonary vasodilator effect. However, the potential role of AZA in the treatment of PH has not been conclusively studied. Therefore, the purpose of the current project is to investigate, the acute hemodynamic clinical effects of AZA in PH patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing RHC for a clinical indication and who are diagnosed with precapillary PH (mPAP ≥25 mmHg, pulmonary wedge pressure (PAWP) ≤15mmHg)

Exclusion Criteria:

* Patients in whom a RHC is clinically not indicated
* pregnant women
* PH in left heart disease or with more than mild chronic obstructive pulmonary disease or restrictive lung disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (PVR) AZA vs. Placebo (rest) | 60 minutes
  At the end of phase at rest
PVR AZA vs. Placebo (exercise) | 60 minutes
  At the end of phase at exercise
PVR AZA vs. Placebo (hypoxia) | 60 minutes
  At the end of phase under hypoxia

SECONDARY OUTCOMES:
partial pressure of the oxygen | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
Oxygen uptake | 15 minutes
minute ventilation | 15 minutes
arterial oxygenation | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
tissue oxygenation | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
mean pulmonary arterial pressure | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
cardiac output | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
cardiac index | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
pulmonary wedge pressure | 60 minutes
  At the end of each phase (rest, exercise and hypoxia)
Borg scale dyspnea and leg effort | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — UniversityHospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duknic M, Lichtblau M, Saxer S, Berlier C, Schneider SR, Schwarz EI, Carta AF, Furian M, Bloch KE, Ulrich S. Comparison of Repetitive Cardiac Output Measurements at Rest and End-Exercise by Direct Fick Using Pulse Oximetry vs. Blood Gases in Patients With Pulmonary Hypertension. Front Med (Lausanne). 2021 Nov 23;8:776956. doi: 10.3389/fmed.2021.776956. eCollection 2021. PMID 34888330